CLINICAL TRIAL: NCT07169591
Title: Exploring the Effect of Hormonal Contraceptives on Postprandial Glucose Handling in Young Healthy Females
Brief Title: Postprandial Glucose Handing in Contraceptive and IUD Users
Acronym: HCPG
Status: Recruiting | Type: Observational
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Kirsten Bell, Principal Investigator, McMaster University
Other Study IDs: 18506
Record Dates: First submitted 2025-08-05; First posted 2025-09-12 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Glucose Homeostasis
Keywords: Glucose; Insulin; Female Health; Hormonal Contraceptive; Intrauterine Device; Oral Contraceptive Pill
MeSH Terms: conditions — Insulin Resistance | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- NAT: Naturally-cycling females
  Interventions: Diagnostic Test: Oral Glucose Tolerance test (75g 2-hour)
- OCP: Combined oral contraceptive users
  Interventions: Diagnostic Test: Oral Glucose Tolerance test (75g 2-hour)
- IUD: Hormonal intrauterine device users
  Interventions: Diagnostic Test: Oral Glucose Tolerance test (75g 2-hour)

INTERVENTIONS:
Diagnostic Test: Oral Glucose Tolerance test (75g 2-hour) — Standard oral glucose tolerance test with blood draws every 15-30 minutes for a 2-hour span

SUMMARY:
Goals: The long-term use of hormonal birth control has been shown to effect glucose handling, or blood sugar regulation, and potentially lead to insulin resistance which increases a person's risk for metabolic diseases such as type 2 diabetes. The goal of this study is to investigate how the body handles glucose, in three groups of young, healthy females: NAT (naturally cycling, or not using hormonal birth control), OCP (taking a birth control pill), and IUD (using an intrauterine device). Objectives: We will investigate if the body's ability to handle glucose differs between these groups. We will also explore if these differences are linked to the levels of primary sex hormones in females, estrogen and progesterone, and if the synthetic versions produced by hormonal birth control have the same negative effect. We will use an oral glucose tolerance test to investigate these potential differences, having participants drink a 75 gram glucose beverage and taking blood samples every 15-30 minutes for a 2-hour timespan. These blood samples will be used to measure glucose and insulin levels in the blood to determine any changes that occur in the body in response to glucose.

DETAILED DESCRIPTION:
Insulin resistance is a common metabolic condition, and is considered a primary risk factor for the development of type 2 diabetes (T2D). As the prevalence of T2D continues to rise, particularly among premenopausal females (18-45 years), it is imperative to conduct additional research in this area. Fluctuations in primary sex hormones in females have been shown to modulate risk for developing impaired glucose tolerance, however, research in this area as well as work investigating synthetic versions of these hormones for OCP and IUD users remains unclear. It is crucial to investigate how hormonal contraceptives can alter glucose tolerance in young, otherwise healthy females, and what downstream effects contraceptives could have later in life.

ELIGIBILITY:
Inclusion Criteria:

* Within 18-45 years
* BMI between 18.5 and 30.0 kg/m2
* Weight stable for the past 6 months (± 2kg)
* VO2peak values within a below average to above average rangea
* Fasting blood glucose <6.0 mMb
* Resting blood pressure <140/90 mmHg

NAT females:

• Regular menstrual cycle for > 6 months (defined as a cycle length of 21-35 days)

OCP users:

* Use of combined OCPs as prescribed for > 3 months
* Second generation levonorgestrel drugs only
* Monophasic formulations only (Alesse, Alysena, Audrina, Aviane, Min-Ovral, Ovima, or Portia)

IUD users:

* Insertion of IUD no fewer than 3 months prior to beginning of study
* Hormonal, levonorgestrel-releasing IUD (Kyleena or Mirena)

Exclusion Criteria:

* Smoking
* Diabetes, cancer, or other metabolic disorders
* Cardiac or gastrointestinal problems
* Infectious disease
* Barium swallow or nuclear medicine scan in the previous 3 weeks
* Pregnant or breastfeeding
* Diagnosis of polycystic ovary syndrome
* Endometriosis
* Use of emergency contraception (e.g., Plan B) within the previous 3 months

NAT females:

• Use of any type of hormonal contraceptive in the previous 3 months

OCP users:

* Not using OCP as prescribed (e.g. missing doses or taking drug inconsistently)
* Use of OCP for longer than 3 years.

IUD users:

* Insertion of Kyleena IUD longer than 2 years.
* Insertion of Mirena IUD longer than 4 years.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We will recruit 54 young healthy recreationally active females (n=18 per group) 18-45 years of age from the following groups: 1) individuals currently taking second generation OCPs containing levonorgestrel, 2) individuals with a levonorgestrel-releasing IUD, and 3) NAT individuals.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Glucose tolerance | 2 hours
  A 2-hour oral glucose tolerance test will be performed in fasted individuals

SECONDARY OUTCOMES:
Glucose and lipid metabolites | Timepoints: 0 minute, 15 minute, 30 minute, 45 minute, 60 minute, 90 minute, 120 minute
  Peak concentration of whole blood glucose
Glucose and lipid metabolites | Timepoints: 0 minute, 15 minute, 30 minute, 45 minute, 60 minute, 90 minute, 120 minute
  Insulin
Glucose and lipid metabolites | Timepoints: 0 minute, 15 minute, 30 minute, 45 minute, 60 minute, 90 minute, 120 minute
  C-peptide
Glucose and lipid metabolites | Fasting (0 min timepoint)
  Concentration of total and high-density lipoprotein cholesterols
Glucose and lipid metabolites | Fasting (0 min timepoint)
  Concentration of non-esterified fatty acids (NEFAs)

OTHER OUTCOMES:
Hormone availability | Fasting (0 min timepoint)
  Concentration of 17b estradiol (endogenous estrogen)
Hormone availability | Fasting (0 min timepoint)
  Concentration of endogenous progesterone
Hormone availability | Fasting (0 min timepoint)
  Concentration of ethinyl estradiol (exogenous estrogen)
Hormone availability | Fasting (0 min timepoint)
  Concentration of levonorgestrel (exogenous progesterone)

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Ivor Wynne Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
To protect participant privacy, IPD will not be available to other researchers.